CLINICAL TRIAL: NCT02445339
Title: Novel Interventions for Alcohol Dependent Frequent Emergency Department Users: Phase IV, Randomized, Open-label, Non-placebo-controlled Study of Extended-release Naltrexone and Care Management on Healthcare Use, Drinking, & Quality of Life
Brief Title: Extended-release Naltrexone and Care Management for Alcohol Dependent Frequent Emergency Department Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-00928; 1K23AA022989-01 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-05-15 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Alcohol Dependence; Alcohol Use Disorder
Keywords: Alcohol Dependence; Alcohol Use Disorder; Care Management; Case Management; Emergency Care Services; Emergency Department; Emergency Room; Extended-release naltrexone; Frequent Users; Health Care Utilization; Medical Management; Naltrexone; Population Health; Public Health; Vivitrol; XR-NTX; XR-NTX+CM; Alcoholism; Alcohol-Related Disorders; Central Nervous System Agents; Chemically-Induced Disorders; Clinical Trial; Emergency Medicine; Mental Disorders; Narcotic Antagonists; Peripheral Nervous System Agents; Pharmacologic Actions; Physiological Effects of Drugs; Sensory System Agents; Substance-Related Disorders
MeSH Terms: conditions — Alcoholism; Emergencies; Patient Acceptance of Health Care; Alcohol-Related Disorders; Chemically-Induced Disorders; Mental Disorders; Substance-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm: XR-NTX+CM (Active Comparator): XR-NTX+CM (Extended Release Naltrexone + Care Management)
  Interventions: Drug: XR-NTX+CM (Extended-Release Naltrexone plus Care Management)
- Standard Care Arm (No Intervention): Standard Care/Alcohol-Medical Management (MM) Only

INTERVENTIONS:
Drug: XR-NTX+CM (Extended-Release Naltrexone plus Care Management) — The intervention arm will receive extended-release naltrexone (XR-NTX) 380mg (4 mL) to be administered as an intramuscular gluteal injection every 28 days up to 12 doses total. Expedited referral to alcohol-medical management. Care Management will include coordination of health care and social services for at least 12 months. Harm-reduction counseling and motivational interviewing to identify and work towards goals. The Standard care arm will receive an expedited alcohol-medical management referral.
  Other Names: Vivitrol
  Arms: Intervention Arm: XR-NTX+CM

SUMMARY:
Our primary aim is to assess the feasibility of initiating treatment in the ED with extended-release naltrexone (XR-NTX) plus care management (CM) vs. standard care and continuing care in cooperation with clinic providers as well as how best to assess outcomes. Secondarily, the investigators will explore its effect on various health outcomes (healthcare utilization and engagement, expenditures, drinking and consequences, quality of life) as well as the association of patient-level characteristics (e.g. sex, race, baseline drinking, health and psychosocial factors, mu opioid receptor genotype) with effectiveness. Determining both how to implement XR-NTX+CM and rigorously test its effects in the ED (phase 1) is essential before planning a large-scale effectiveness trial (phase 2).

DETAILED DESCRIPTION:
Aim #1: To conduct a feasibility and acceptability study of XR-NTX+CM treatment in alcohol dependent patients with frequent ED use.

Hypothesis: Enrollment of a limited number of subjects will allow identification of optimal processes for a definitive trial.

Aim #2: To conduct an analysis of the effect of this intervention on healthcare utilization and engagement, drinking outcomes, quality of life, and consequences of drinking (initial analysis will be exploratory).

Hypothesis: Measuring changes in healthcare utilization, drinking metrics, and indicators of quality of life and consequences will provide preliminary data on intervention effect size on various outcomes of interest to inform the second phase, definitive trial.

Aim #3: To identify patient-level characteristics associated with effectiveness.

Hypothesis: Exploratory analysis of patient and system-level characteristics possibly associated with effectiveness will inform treatment choice to maximize the probability of successful outcome. Factors assessed will include data collected in ongoing investigations of pharmacotherapy for alcohol dependence, including mu opioid receptor (OPRM1) genotypes, to facilitate comparison across study populations and settings.

This a phase IV, randomized, open-label, non-placebo-controlled, single-center study of the feasibility, acceptability, and effect of initiating treatment in the ED with extended-release naltrexone 380mg intramuscular injection compared to standard care in subjects with severe alcohol use disorders (i.e. alcohol dependence) and frequent emergency department use. In the first two years, we will finalize study preparations, recruit and randomize 50 subjects for the pilot phase of this study. The duration of each subject's participation will be 12 months. Thereafter, in the second phase of study, we will enroll an additional 250 subjects (for a total of 300 subjects) to address remaining feasibility and acceptability concerns and test effects.

The study investigators (PI and RA) will collect process data, including barriers and facilitators encountered in the completion of all study procedures. For the following study procedures, study investigators (the PI and RAs) will enter data directly into New York University Langone Medical Center (NYULMC) internal REDCap system for use on portable tablet computers.

Synopsis of Study Procedures:

The following study procedures are described in greater detail elsewhere in this protocol.

Patients will be prescreened for potential eligibility and added to an automated alert system linked to ED registration by Bellevue Care Managers as part of an ongoing quality improvement initiative. When a potentially eligible patient presents to the ED, an automated page will be delivered to the study PI and Bellevue ED social work and care management staff, prompting consultation and potential referral of the patient to study investigators (PI/RA) for recruitment (See 4.3 Subject Recruitment and Screening). ED medical providers (inclusive of ED physicians, nurses, social workers, and care managers) will notify study investigators (PI/RA) when potentially eligible patients are present in the ED. The medical provider will introduce the PI/RA to clinically sober and medically stable patients who have given their permission to be approached. The PI/RA will describe the study, confirm capacity to consent using the University of California San Diego Brief Assessment of Capacity to Consent to Research (UBACC), and obtain written informed consent. The PI/RA will confirm eligibility by performing a chart and laboratory review (liver enzymes, pregnancy, urine drug screen), history and examination, and diagnostic interview to confirm alcohol dependence and assess for opioid use and chronic pain. The PI/RA will conduct research intake assessments and interview and collect blood for biomarker (5mL) and genetic (10mL) analyses. The PI/RA will randomize subjects to intervention (XR-NTX+CM) or Standard Care using a random number generator with randomly permuted blocks with allocations contained within opaque sealed envelopes.

1. For subjects randomized to the Intervention Arm, the PI/RA will confirm the drug screen is negative for opioids prior to administering XR-NTX 380mg as an intramuscular gluteal injection. The PI/RA will facilitate a person-centered, harm-reduction-based motivational interview, , and psychosocial assessment/interview to inform subjects' care-management plans. Subjects will receive a one-week referral to Bellevue ambulatory care for initial Alcohol-Medical Management (MM) and will also be scheduled every 4 weeks (after most recent XR-NTX injection) for MM and XR-NTX injections. When possible, participants who miss MM-injection visits will be navigated to clinic upon their next ED presentation and/or may receive MM and XR-NTX in the ED. XR-NTX will be administered by the PI or a provider (physician, physician assistant, or registered nurse) who is trained in the administration of XR-NTX. The schedule for MM-Injection visits is weeks 4, 8, 12, 16, 20, and 24. Participants may be offered to continue XR-NTX treatment through this study for as many has 12 injections in total as we explore the feasibility, acceptability and potential benefits of extending treatment duration to 12 months. The schedule for potential additional MM-Injection visits is weeks 28, 32, 36, 40, and 44. Research assessment visits will occur at weeks 12, 24, and 48 and may be conducted up to 28 days prior to- or 90 days after- date in which research visits are due. During research visits, the PI/RA will repeat the assessments that were conducted at the initial enrollment visit plus adverse events and participant satisfaction and we will collect a 5mL blood sample to examine alcohol consumption biomarkers. Subject participation ends after the week-48 research visit.
2. For subjects randomized to the Standard care arm, the PI/RA will provide referral to Bellevue ambulatory care for MM without further intervention. Research assessment visits will occur at weeks 12, 24, and 48 and may be conducted up to 28 days prior to- or 90 days after- date in which research visits are due. During research visits, the PI/RA will repeat the assessments that were conducted at the initial enrollment visit plus adverse events and participant satisfaction and we will collect a 5mL blood sample to examine alcohol consumption biomarkers. Subject participation ends after the week-48 research visit.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be eligible for study enrollment:

1. English or Spanish speaking*

   *Non-English Spanish speaking patients will not be enrolled initially until study documents have been translated, back translated, and approved by the Institutional Review Board (IRB).
2. Emergency Department patient
3. Aged 18-80
4. Have had >4 emergency department visits within 12 months for 2 consecutive 12-month periods. Period of time can be extended by up to 6 months if incarcerated or institutionalized for ≥ 6 months.
5. Meet Diagnostic and Statistical Manual version IV (DSM-IV) criteria for alcohol dependence or & DSM-V criteria for alcohol use disorder, severe.
6. Have ≥2 days/week of heavy drinking (>4 drinks/day)
7. Capable of giving informed consent.

Exclusion Criteria

Subjects who meet any of the following criteria will be ineligible for study enrollment:

1. Active opioid dependence
2. Acute or chronic pain requiring opioid treatment
3. Acute liver injury (liver aminotransferase concentrations >5 times the upper limit of normal)
4. Health condition considered unsafe for inclusion (at discretion of PI and/or attending physician)
5. Lack of capacity or willingness to consent
6. Currently prescribed pharmacotherapy for alcohol dependence (not including treatment of acute alcohol withdrawal syndrome)
7. Previous significant adverse reaction to naltrexone or diluent
8. Pregnant, nursing, or not using effective methods of birth control
9. Prisoners (as defined by Office of Human Research Protection) at the time of enrollment ARE NOT ELIGIBLE for study entry. However, subjects who become prisoners after being enrolled will be included and not be withdrawn from the study. Patients on parole or probation are eligible for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P McCormack, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Bellevue Hospital Center, New York, New York, United States

REFERENCES:
- [Background] McCormack RP, Williams AR, Goldfrank LR, Caplan AL, Ross S, Rotrosen J. Commitment to assessment and treatment: comprehensive care for patients gravely disabled by alcohol use disorders. Lancet. 2013 Sep 14;382(9896):995-7. doi: 10.1016/S0140-6736(12)62206-5. Epub 2013 Apr 19. No abstract available. PMID 23602314
- [Background] McCormack RP, Hoffman LF, Wall SP, Goldfrank LR. Resource-limited, collaborative pilot intervention for chronically homeless, alcohol-dependent frequent emergency department users. Am J Public Health. 2013 Dec;103 Suppl 2(Suppl 2):S221-4. doi: 10.2105/AJPH.2013.301373. Epub 2013 Oct 22. PMID 24148034
- [Background] McCormack RP, Hoffman LF, Norman M, Goldfrank LR, Norman EM. Voices of homeless alcoholics who frequent Bellevue Hospital: a qualitative study. Ann Emerg Med. 2015 Feb;65(2):178-86.e6. doi: 10.1016/j.annemergmed.2014.05.025. Epub 2014 Jun 26. PMID 24976534
- [Background] McCormack RP, Gallagher T, Goldfrank LR, Caplan AL. Including frequent emergency department users with severe alcohol use disorders in research: assessing capacity. Ann Emerg Med. 2015 Feb;65(2):172-7.e1. doi: 10.1016/j.annemergmed.2014.09.027. Epub 2014 Oct 23. PMID 25447556
- [Background] Hamilton BH, Sheth A, McCormack RT, McCormack RP. Imaging of frequent emergency department users with alcohol use disorders. J Emerg Med. 2014 Apr;46(4):582-7. doi: 10.1016/j.jemermed.2013.08.129. Epub 2014 Jan 10. PMID 24412058
- [Background] Lee JD, Grossman E, DiRocco D, Truncali A, Hanley K, Stevens D, Rotrosen J, Gourevitch MN. Extended-release naltrexone for treatment of alcohol dependence in primary care. J Subst Abuse Treat. 2010 Jul;39(1):14-21. doi: 10.1016/j.jsat.2010.03.005. Epub 2010 Apr 2. PMID 20363090
- [Background] Collins SE, Saxon AJ, Duncan MH, Smart BF, Merrill JO, Malone DK, Jackson TR, Clifasefi SL, Joesch J, Ries RK. Harm reduction with pharmacotherapy for homeless people with alcohol dependence: protocol for a randomized controlled trial. Contemp Clin Trials. 2014 Jul;38(2):221-34. doi: 10.1016/j.cct.2014.05.008. Epub 2014 May 17. PMID 24846619

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Started | 25 | 25
Completed | 13 | 10
Not Completed | 12 | 15
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.3) | 54.2 (8.6) | 55 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 6 | 6 | 12
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Heavy Drinking Days
Description: Self-reported
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
days | 62 (9.4) | 0 (0)

2. Secondary Outcome: Number of Heavy Drinking Days
Description: Self-reported
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
days | 32 (9.1) | 25 (7.9)

3. Secondary Outcome: Number of Heavy Drinking Days
Description: Self-reported
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
days | 0 (0) | 37 (9.5)

4. Secondary Outcome: Short Inventory of Problems Related to Alcohol (SIP-2R) Score
Description: SIP-2R is a measure for assessing recent adverse consequences associated with alcohol use. SIP-2R consists of 15 events that are scored from 0 (never) to 3 (daily or almost daily). The total score range is 0-45; the higher the score, the more problems related to alcohol use.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 25.4 (10.6) | 24.9 (13.2)

5. Secondary Outcome: Short Inventory of Problems Related to Alcohol (SIP-2R) Score
Description: as for outcome 4
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 20.8 (14.6) | 25.3 (15)

6. Secondary Outcome: Short Inventory of Problems Related to Alcohol (SIP-2R) Score
Description: as for outcome 4
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 13.1 (11) | 17.1 (15)

7. Secondary Outcome: Carbohydrate-deficient Transferrin (CDT) Levels
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: %CDT
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
%CDT | 5.4 (4.6) | 2.8 (2.8)

8. Secondary Outcome: Carbohydrate-deficient Transferrin (CDT) Levels
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: %CDT
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
%CDT | 3.5 (3.4) | 4.7 (4.3)

9. Secondary Outcome: Carbohydrate-deficient Transferrin (CDT) Levels
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: %CDT
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
%CDT | 2.6 (2.1) | 3.7 (3)

10. Secondary Outcome: Gamma-glutamyl Transferase (GGT) Levels
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
units/liter | 197.8 (290) | 107.8 (136.8)

11. Secondary Outcome: Gamma-glutamyl Transferase (GGT) Levels
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
units/liter | 154.8 (305.6) | 146.8 (193.2)

12. Secondary Outcome: Gamma-glutamyl Transferase (GGT) Levels
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
units/liter | 111.8 (178.2) | 109.3 (139)

13. Secondary Outcome: EuroQoL-5 Dimensions (EQ-5D) Score
Description: EQ-5D is a standardized measure of health-related quality of life. A visual analogue scale is used to record an individual's valuation of defined EQ-5D profiles. The total score range is 0-100; the higher the score, the better the health state (0=worst imaginable health state, 100=best imaginable health state).
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 67.1 (25.2) | 56.1 (25.3)

14. Secondary Outcome: EuroQoL-5 Dimensions (EQ-5D) Score
Description: as for outcome 13
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 70.4 (19.8) | 68.8 (19.8)

15. Secondary Outcome: EuroQoL-5 Dimensions (EQ-5D) Score
Description: as for outcome 13
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
Number analyzed (Participants) | 13 | 10
score on a scale | 77.6 (14.1) | 56.7 (23.9)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: During research visits in the Emergency Department (ED), the PI/RA will collect adverse event information.
Arm/Group | Intervention Arm: XR-NTX+CM | Standard Care Arm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02445339/Prot_SAP_000.pdf